CLINICAL TRIAL: NCT05978232
Title: Prospective Pilot Study of Navigator-Assisted Hypofractionation (NAVAH) Impact on Radiation Therapy Completion in Black Breast & Prostate Cancer Patients
Brief Title: NAVAH Impact on Radiation Therapy Completion in Black Breast & Prostate Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Gilead Sciences (Industry); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1123
Record Dates: First submitted 2023-06-06; First posted 2023-08-07 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: Radiation Therapy; Navigator-Assisted Hypofractionation
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Navigator-Assisted Hypofractionation (NAVAH) (Experimental): This pilot cohort study is designed as follows:
  1. Navigator discussion with patients prior to the start of radiation therapy simulation (15-30 minutes).
  2. Navigator administration of survey with patients after completion of radiation therapy simulation but before the start of radiation therapy (30-45 minutes)
  3. Navigator administration of post-treatment survey and financial toxicity survey instrument after the completion of radiation therapy (60 minutes).
  Interventions: Behavioral: NAVAH

INTERVENTIONS:
Behavioral: NAVAH — Patient navigator program that aims to inform African-American prostate and breast cancer patients about their treatment options, specifically radiotherapy

SUMMARY:
African-Americans have disparately limited access to optimal cancer care. They have the highest overall cancer death rate and shortest survival time of any racial or ethnic group in the United States. Elucidation of disparities in access to cancer care are important since previous work has indicated that when equal access to RT in Radiation Therapy Oncology Group (RTOG) prospective randomized trials is granted, race does not independently affect outcomes, a finding similar to work conducted in Level I evidence-proven optimal management of curable neurologic conditions. Breast cancer is the most common cancer in African-American women and Prostate cancer is the most common cancer in African-American men. African-American breast & prostate cancer participants are less likely to receive standard-of-care radiation therapy.

Previous work has identified that compared to Caucasian women with breast cancer, African-American women are 48% more likely to have RT omission during treatment, 167% less likely to receive timely completion of RT after breast-conserving surgery, 40% less likely to complete RT, and significantly more likely to experience RT treatment delays. Shorter course radiation therapy may reduce disparities in radiation therapy care facing African-American breast cancer participants.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed Breast or Prostate Cancer.
* Subjects must be Age >18 years. This study requires informed consent by the subject; as children are not able to perform this without parental approval, subjects < age 18 are excluded from this study.
* Subjects must be of African - American race.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects NOT of African - American ethnicity.
* Subjects WITHOUT histologically or cytologically confirmed Breast or Prostate Cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of barriers to navigator access | Immediately following radiotherapy treatment
  Survey-based methods will be used to assess barriers facing under-represented minority cancer patient access to patient navigation. This study will use a patient-completed, culturally sensitive survey adapted from "Walking Forward," a patient navigator program providing culturally appropriate community education on cancer, screening and treatment, to include barriers to specific RT regimens, and concerns regarding transportation.

SECONDARY OUTCOMES:
Assess the impact of patient navigation on patient access to radiation oncology care | Immediately following radiotherapy treatment
  Qualitative mechanisms will be used to assess the impact of patient navigation on patient access to radiation oncology care and consequently utilization of standard of care modalities. This study will use patient-completed surveys to evaluate the impact of patient navigation on access to short-course RT by using a culturally sensitive survey adapted from "Walking Forward", a patient navigator program providing culturally appropriate community education on cancer, screening and treatmen. The feedback provided by patients on the impact of patient navigation will be compared- before and after RT, and will also be compared against feedback from patients who did not received patient navigation.
Minority financial toxicity differences | Immediately following radiotherapy treatment
  This study will use patient-completed surveys to evaluate the impact of financial hardship in African-American breast cancer patients. Patient scores from an evidence-based tool, "The COmprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy (COST-FACIT)" will be used to compare financial hardship in each group of patients with early-stage breast cancer who have received a lumpectomy. Surveys will investigate differences in financial toxicity survery scores experienced by underrepresented minorities receiving conventional versus short-course RT.

CONTACTS AND LOCATIONS:
Overall Officials: Shearwood McClelland III, MD, Principal Investigator — University Hospitals Cleveland Medical Center Seidman Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] McClelland S 3rd, Burnette U, Onyewadume L, Smith TK, Speers CW. Impact of Patient Navigation on Radiation Therapy Completion in Black Breast Cancer Patients: Early Phase I Trial Results From the Navigator-Assisted Hypofractionation (NAVAH) Program. Am J Clin Oncol. 2025 Oct 15. doi: 10.1097/COC.0000000000001257. Online ahead of print. PMID 41091946
- [Derived] Posani S, Burnette UJ, McClelland S 3rd. Quantification of Postdiagnosis Cancer Patient Navigation. Am J Clin Oncol. 2025 Dec 1;48(12):610-613. doi: 10.1097/COC.0000000000001225. Epub 2025 Jun 17. PMID 40525892
- [Derived] Davis KJ, Burnette UJ, Sun Y, Stephens MJ, Onyewadume L, McClelland S 3rd. Medical Racism and Physician Trust Impressions of African-American Breast Cancer Patients Enrolled on the Navigator-Assisted Hypofractionation (NAVAH) Phase I Clinical Trial. Am J Clin Oncol. 2025 Jul 1;48(7):339-341. doi: 10.1097/COC.0000000000001183. Epub 2025 Mar 3. PMID 40025854